CLINICAL TRIAL: NCT02523131
Title: An Open-label, Multi-centre, Randomised, Single-period, Parallel Design Study to Assess the Efficacy, Safety, Utility and Psychosocial Effect of 12 Week Day and Night Automated Closed Loop Glucose Control Combined With Pump Suspend Feature Compared to Sensor Augmented Insulin Pump Therapy in Youth and Adults With Type 1 Diabetes With Sub-optimal Glucose Control Under Free Living Conditions
Brief Title: Home Testing of Day and Night Closed Loop With Pump Suspend Feature
Acronym: APCam11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Jaeb Center for Health Research (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); International Diabetes Center at Park Nicollet (Other); University of Colorado, Denver (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APCam11
Record Dates: First submitted 2015-08-09; First posted 2015-08-14 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases
Keywords: Type 1 diabetes; Closed-loop glucose control; Artificial Pancreas; Continuous subcutaneous insulin infusion; Continuous glucose monitoring; threshold suspend; predictive low glucose suspend
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24/7 closed loop insulin delivery (Experimental): Unsupervised home use of day and night automated closed loop insulin delivery system (FlorenceM) combined with pump suspend feature over a 12-week period using 24/7 Medtronic insulin pump 640G and Android smartphone.
  Interventions: Device: FlorenceM
- Sensor augmented pump therapy (Active Comparator): Insulin pump therapy combined with unmasked real-time continuous glucose monitoring system for 12 weeks using Medtronic insulin pump 640G. Pump suspend features will be turned off.
  Interventions: Device: Medtronic insulin pump 640G

INTERVENTIONS:
Device: FlorenceM — The automated closed loop system (FlorenceM) will consist of:
  * Next generation sensor augmented Medtronic insulin pump 640G (Medtronic Minimed, CA, USA) incorporating the Medtronic Enlite 3 family real time CGM and glucose suspend feature.
  * An Android smartphone containing the Cambridge model predictive algorithm and communicating wirelessly with the insulin pump using a proprietary translator device.
  Arms: 24/7 closed loop insulin delivery
Device: Medtronic insulin pump 640G — Next generation sensor-augmented Medtronic insulin pump 640G (Medtronic Minimed, CA, USA) incorporating the Medtronic Enlite 3 family real time CGM. Glucose suspend features will be turned off.
  Arms: Sensor augmented pump therapy

SUMMARY:
The main study objective is to determine whether day and night automated closed loop glucose control combined with pump suspend feature will improve glucose control and reduce the burden of hypoglycaemia compared to sensor augmented insulin pump therapy alone.

This is an open-label, multi-centre, multi-national, single-period, randomised, parallel group design study, involving a three-month period of home study during which day and night glucose levels will be controlled either by a closed loop system combined with pump suspend feature (intervention group) or by sensor augmented insulin pump therapy (control group).

It is expected that up to 100 subjects, aiming for 84 randomised subjects [42 youth (6 to 21 years), and 42 adults (22 years and older)], with type 1 diabetes will be recruited through paediatric and adult outpatient diabetes clinics in each of the investigation centres. Subjects who drop out within the first four weeks of the intervention may be replaced. Participants will all be on subcutaneous insulin pump therapy and will have proven competencies both in the use of the study insulin pump and the study CGM device.

Subjects in the intervention group will receive appropriate training in the safe use of closed loop insulin delivery system and pump suspend feature. All subjects will have regular contact with the study team during the home study phase including 24/7 telephone support. The primary outcome is between group differences in the time spent in the target glucose range from 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on CGM glucose levels during the 12 week free living phase. Secondary outcomes are HbA1 at the end of treatment period, the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Safety evaluation comprises assessment of the frequency of severe hypoglycaemic episodes.

DETAILED DESCRIPTION:
Purpose of the study:

To determine whether day and night automated closed loop glucose control combined with pump suspend feature will improve glucose control as measured by glycated haemoglobin and reduce the burden of hypoglycaemia compared to sensor augmented insulin pump therapy.

Study objectives:

1. EFFICACY: The objective is to assess efficacy of day and night automated closed loop glucose control combined with pump suspend feature in maintaining glucose levels within the target range from 3.9 to 10.0mmol/l (70 to 180mg/dl) based on subcutaneous continuous glucose monitoring (CGM), as compared to sensor augmented insulin pump therapy.
2. SAFETY: The objective is to evaluate the safety of day and night automated closed loop glucose control combined with pump suspend feature, in terms of episodes of severe hypoglycaemia and other adverse events.
3. UTILITY: The objective is to determine the frequency and duration of the use of the automated closed loop system.
4. PSYCHOSOCIAL: Subjects' and family members' perception in terms of life-style change, diabetes management and fear of hypoglycaemia will be assessed using validated questionnaires and semi-structured qualitative interviews. Cognitive functions will be assessed using validated computerized cognitive tests.

Study design:

An open-label, multi-centre, multi-national, randomised, single-period, parallel group study, contrasting day and night automated closed loop glucose control combined with pump suspend feature with sensor augmented insulin pump therapy

Population:

84 participants randomised (42 youth and 42 adults). Each centre will aim to recruit between 05 and 20 participants.

Maximum duration of study for a subject :

18 weeks

Recruitment:

The subjects will be recruited through the paediatric and adult diabetes outpatient clinics at each centre.

Consent:

Written consent/assent will be obtained from participants and/or guardians according to REC/IRB requirements.

Screening assessment:

Eligible participants will undergo a screening evaluation where blood samples for full blood count, renal, liver, thyroid function and anti-transglutaminase antibodies with IgA levels will be taken (if not done in the previous 3 months). Random C-peptide, glucose and HbA1c will also be measured, and a urine pregnancy test in females of child-bearing potential.

Questionnaires investigating participants' quality of life, psychosocial functioning and response to their current treatment will be distributed. Cognitive assessment will be made using validated computerized cognitive tests.

Study Training:

Training sessions on the use of study CGM, insulin pump (and closed loop system for those randomised to the intervention group) will be provided by the research team. Training session on the use of real-time CGM and on how to interpret real-time and retrospective stored data will be provided to all subjects/carers using written material.

Run-in Period:

During a 4 week run-in period, subjects will use study CGM and insulin pump. The research team will contact subject once weekly during the run-in period, and subjects will also be able to contact the research team for support and treatment optimisation as necessary. For compliance and to assess the ability of the subject to use the CGM and study pump safely, at least 12 days of CGM data need to be recorded and safe use of study insulin pump demonstrated during the last 14 days of run-in period.

Competency assessment:

Competency on the use of study insulin pump and study CGM will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required.

Randomisation:

Eligible subjects will be randomised using randomisation software to the use of real-time CGM and pump suspend feature combined with day and night closed loop or to sensor augmented insulin pump therapy.

1. Automated day and night closed loop insulin delivery (intervention arm) combined with pump suspend feature (interventional arm):

   At the start, a blood sample will be taken for the measurement of HbA1c and a urine pregnancy test in females of child-bearing potential.

   A subset of participants will be interviewed to enable their historical diabetes management practices, everyday work and family lives, and their initial expectations of using closed loop technology to be captured and explored in-depth.

   Subjects will be admitted to the clinical facility on Day 1. Training on the use of closed loop and pump suspend feature will be provided by the research team. During the next 2-4 hours patient will operate the system under the supervision of the clinical team. Competency on the use of closed loop system will be evaluated. Subjects will use closed loop and pump suspend feature for 12 weeks.
2. Sensor augmented insulin pump therapy (control arm):

A blood sample will be taken for the measurement of HbA1c and a urine pregnancy test in females of child-bearing potential. Subjects will use sensor augmented insulin pump therapy without pump suspend feature for 12 weeks.

End of study assessments:

* A blood sample will be taken for measurement of HbA1c.
* Validated questionnaires evaluating the impact of the devices employed on life change, diabetes management will be completed.
* Cognitive assessment will be made using validated computerized cognitive tests.
* Follow-up interviews will be undertaken with the subset of participants/family members at the end of the closed loop intervention.

Procedures for safety monitoring during trial:

* Standard operating procedures for monitoring and reporting of all adverse events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.
* Subjects will be asked to test and record blood or urine ketones if their finger prick glucose is above 14.0mmol/l (250mg/dl) in the morning on waking, as part of the safety assessment for hyperglycaemia.
* A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of patients on safety grounds:

A subject, parent, or guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

1. Serious adverse events
2. Significant protocol violation or non-compliance
3. Failure to satisfy competency assessment
4. Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest
5. Pregnancy, planned pregnancy, or breast feeding
6. Allergic reaction to insulin
7. Technical grounds (e.g. subject relocates)

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 6 years or older [with equal proportion of youth (6 to 21 years) and adults (22 years and older)]
2. The subject has type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
3. The subject will have been an insulin pump user for at least 3 months, with good knowledge of insulin self-adjustment as judged by the investigator
4. The subject is treated with one of the rapid acting insulin analogues (insulin Aspart, Lispro or Glulisine)
5. The subject is willing to perform regular capillary blood glucose monitoring, with at least 4 blood glucose measurements taken every day
6. Screening HbA1c ≥ 7.5% (58.5mmol/mol) and ≤ 10 % (86mmol/mol) based on analysis from local laboratory or equivalent [with equal proportion of subjects above and below HbA1c 8.5% (69mmol/mol)]
7. The subject is literate in English
8. The subject is willing to wear glucose sensor
9. The subject is willing to wear closed loop system at home
10. The subject is willing to follow study specific instructions
11. The subject is willing to upload pump and CGM data at regular intervals
12. The subject is willing to restrict alcohol consumption to ≤ 2 units per day throughout the study period
13. Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening.
14. The subject lives with someone who is trained to administer intramuscular glucagon and is able to seek emergency assistance.
15. The subject has access to WIFi at home.

Exclusion Criteria:

1. Non-type 1 diabetes mellitus including those secondary to chronic disease
2. Subject using real-time CGM on regular basis in preceding 3 months
3. Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
4. Untreated coeliac disease or thyroid disease or subject is being treated for hypothyroidism at time of screening
5. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, non-selective beta-blockers and MAO inhibitors etc.
6. Known or suspected allergy to insulin
7. Subjects with clinically significant nephropathy (eGFR < 45ml/min) or on dialysis, neuropathy or active retinopathy (defined as presence of maculopathy or proliferative changes) as judged by the investigator
8. Adults: one or more episodes of severe hypoglycaemia as defined by American Diabetes Association (33) in preceding 6 months; Youth: recurrent incidents of severe hypoglycaemia during the previous 6 months (Adults and adolescents: severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions including episodes of hypoglycaemia severe enough to cause unconsciousness, seizures or attendance at hospital; children: severe hypoglycaemia is defined as an event associated with a seizure or loss of consciousness);
9. Random C-peptide > 100pmol/l with concomitant plasma glucose >4 mmol/l (72 mg/dl)
10. Regular use of acetaminophen
11. Lack of reliable telephone facility for contact
12. Total daily insulin dose ≥ 2 IU/kg/day
13. Total daily insulin dose < 15 IU/day
14. Pregnancy, planned pregnancy, or breast feeding
15. Severe visual impairment
16. Severe hearing impairment
17. Significantly reduced hypoglycaemia awareness in subjects 18 year and older (screening Gold score > 4)
18. Subjects using implanted internal pace-maker
19. Patients with medically documented allergy towards the adhesive (glue) of plasters or Subject is unable to tolerate tape adhesive in the area of sensor placement
20. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which potentially are possible to be used for localisation of the glucose sensor)
21. Subject is currently abusing illicit drugs
22. Subject is currently abusing prescription drugs
23. Subject is currently abusing alcohol
24. Subject is using pramlintide (Symlin) at time of screening
25. Subject has elective surgery planned that requires general anaesthesia during the course of the study
26. Subject is a shift worker with working hours between 10pm and 8am
27. Subject has a sickle cell disease, haemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
28. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
29. Subject diagnosed with current eating disorder such as anorexia or bulimia
30. Subject plans to use significant quantity of herbal preparations (use of over the counter herbal preparation for 30 consecutive days or longer period during the study) or significant quantity of vitamin supplements (four times the recommended daily allowance used for 30 consecutive days or longer period during the study) during the course of their participation in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range from 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on CGM glucose levels | 12 week intervention phase
  both arms

SECONDARY OUTCOMES:
HbA1c at the end of treatment period | HbA1c will be taken at the end of 12-week study intervention.
  Between group differences in HbA1c levels at the end of treatment period adjusted for pre-study period HbA1c level.
Time spent below target glucose (3.9mmol/l)(70mg/dl) | 12 week intervention phase
  both arms
Time spent above target glucose (10.0 mmol/l) (180 mg/dl) | 12 week intervention phase
  both arms
Average of glucose levels | 12 week intervention phase
  both arms
The time with glucose levels < 3.5 mmol/l (63mg/dl) and <2.8 mmol/l (50mg/dl) | 12 week intervention phase
  both arms
The time with glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l) (300mg/dl) | 12 week intervention phase
  both arms
Total, basal and bolus insulin dose | 12 week intervention phase
  both arms
AUC of glucose below 3.5mmol/l (63mg/dl) | 12 week intervention phase
  both arms
Standard deviation of glucose levels | 12 week intervention phase
  both arms
Coefficient of variation of glucose levels | 12 week intervention phase
  both arms
Number of pump suspend events | 12 week intervention phase
  closed-loop arm only
Change of body weight from screening to end of study | 12 week intervention phase
  both arms

OTHER OUTCOMES:
Number of episodes of severe hypoglycaemia per subject and incidence rate per 100-person years | 12 week intervention phase
  Comparison of safety outcomes between the two treatment groups only include those events occurring on or after randomization until the last visit date or the last event date (whichever is later).
Number of subjects with severe hypoglycemia events | 12 week intervention phase
  Comparison of safety outcomes between the two treatment groups only include those events occurring on or after randomization until the last visit date or the last event date (whichever is later).
Number of subjects with severe hyperglycemia events as defined by fingerprick glucose >16.7 mmol/l (>300 mg/dl) and plasma ketones >0.6 mmol/l | 12 week intervention phase
  Comparison of safety outcomes between the two treatment groups only include those events occurring on or after randomization until the last visit date or the last event date (whichever is later).
Number of subjects with DKA events | 12 week intervention phase
  Comparison of safety outcomes between the two treatment groups only include those events occurring on or after randomization until the last visit date or the last event date (whichever is later).
Number of any other serious adverse event reported | 12 week intervention phase
  Comparison of safety outcomes between the two treatment groups only include those events occurring on or after randomization until the last visit date or the last event date (whichever is later).
Amount of CL system use | 12 week intervention phase
  Utility evaluation. The amount of system use in the CL arm will be calculated over the period starting from the day after treatment initiation until the earlier of the 12 week visit date or Day 84 from randomization (whichever comes first).
Amount of CGM use | 12 week intervention phase
  Utility evaluation. The amount of CGM use in both arm will be calculated over the period starting from the day after treatment initiation until the earlier of the 12 week visit date or Day 84 from randomization (whichever comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — Department of Paedatrics, University of Cambridge, UK; David B Dunger, Prof, Principal Investigator — Department of Paedatrics, University of Cambridge, UK; Fiona Campbell, MD, Principal Investigator — St James's University Hospital, Leeds, UK; Amy Criego, Prof, Principal Investigator — International Diabetes Center at Park Nicollet, Minneapolis, USA; Mark Evans, MD, Principal Investigator — Wellcome Trust-MRC Institute of Metabolic Science, University of Cambridge, Cambridge, UK; Lalantha Leelarathna, PhD, Principal Investigator — Manchester Diabetes Centre, Manchester Royal Infirmary, Manchester, UK; Richard Bergenstal, Prof, Principal Investigator — International Diabetes Center at Park Nicollet, Minneapolis, USA; Viral Shah, MD, Principal Investigator — Barbara Davis Center for Childhood Diabetes, Aurora, USA; Daniela Elleri, MD, Principal Investigator — Endocrine/Diabetes Department, Royal Hospital for Sick Children, Edinburgh, UK
Locations (8):
- United States (3):
  - University of Colorado Denver, Aurora, Colorado
  - International Diabetes Center at Park Nicollet, Minneapolis, Minnesota
  - International Diabetes Centre at Park Nicollet, Minneapolis, Minnesota
- United Kingdom (5):
  - University of Cambridge, Cambridge
  - Wellcome Trust-MRC Institute of Metabolic Science, Cambridge
  - Royal Hospital for Sick Children, Edinburgh
  - Leeds Teaching Hospitals, Leeds
  - Manchester Diabetes Centre, Manchester Royal Infirmary, Manchester

REFERENCES:
- [Background] Hovorka R. Artificial Pancreas Project at Cambridge 2013. Diabet Med. 2015 Aug;32(8):987-92. doi: 10.1111/dme.12766. Epub 2015 Apr 15. PMID 25819473
- [Background] Leelarathna L, Dellweg S, Mader JK, Allen JM, Benesch C, Doll W, Ellmerer M, Hartnell S, Heinemann L, Kojzar H, Michalewski L, Nodale M, Thabit H, Wilinska ME, Pieber TR, Arnolds S, Evans ML, Hovorka R; AP@home Consortium. Day and night home closed-loop insulin delivery in adults with type 1 diabetes: three-center randomized crossover study. Diabetes Care. 2014 Jul;37(7):1931-7. doi: 10.2337/dc13-2911. PMID 24963110
- [Background] Thabit H, Lubina-Solomon A, Stadler M, Leelarathna L, Walkinshaw E, Pernet A, Allen JM, Iqbal A, Choudhary P, Kumareswaran K, Nodale M, Nisbet C, Wilinska ME, Barnard KD, Dunger DB, Heller SR, Amiel SA, Evans ML, Hovorka R. Home use of closed-loop insulin delivery for overnight glucose control in adults with type 1 diabetes: a 4-week, multicentre, randomised crossover study. Lancet Diabetes Endocrinol. 2014 Sep;2(9):701-9. doi: 10.1016/S2213-8587(14)70114-7. Epub 2014 Jun 16. PMID 24943065
- [Background] Hovorka R, Elleri D, Thabit H, Allen JM, Leelarathna L, El-Khairi R, Kumareswaran K, Caldwell K, Calhoun P, Kollman C, Murphy HR, Acerini CL, Wilinska ME, Nodale M, Dunger DB. Overnight closed-loop insulin delivery in young people with type 1 diabetes: a free-living, randomized clinical trial. Diabetes Care. 2014;37(5):1204-11. doi: 10.2337/dc13-2644. PMID 24757227
- [Derived] Lawton J, Blackburn M, Breckenridge JP, Hallowell N, Farrington C, Rankin D. Ambassadors of hope, research pioneers and agents of change-individuals' expectations and experiences of taking part in a randomised trial of an innovative health technology: longitudinal qualitative study. Trials. 2019 May 27;20(1):289. doi: 10.1186/s13063-019-3373-9. PMID 31133076
- [Derived] Tauschmann M, Thabit H, Bally L, Allen JM, Hartnell S, Wilinska ME, Ruan Y, Sibayan J, Kollman C, Cheng P, Beck RW, Acerini CL, Evans ML, Dunger DB, Elleri D, Campbell F, Bergenstal RM, Criego A, Shah VN, Leelarathna L, Hovorka R; APCam11 Consortium. Closed-loop insulin delivery in suboptimally controlled type 1 diabetes: a multicentre, 12-week randomised trial. Lancet. 2018 Oct 13;392(10155):1321-1329. doi: 10.1016/S0140-6736(18)31947-0. Epub 2018 Oct 3. PMID 30292578
- [Derived] Bally L, Thabit H, Tauschmann M, Allen JM, Hartnell S, Wilinska ME, Exall J, Huegel V, Sibayan J, Borgman S, Cheng P, Blackburn M, Lawton J, Elleri D, Leelarathna L, Acerini CL, Campbell F, Shah VN, Criego A, Evans ML, Dunger DB, Kollman C, Bergenstal RM, Hovorka R. Assessing the effectiveness of a 3-month day-and-night home closed-loop control combined with pump suspend feature compared with sensor-augmented pump therapy in youths and adults with suboptimally controlled type 1 diabetes: a randomised parallel study protocol. BMJ Open. 2017 Jul 13;7(7):e016738. doi: 10.1136/bmjopen-2017-016738. PMID 28710224